CLINICAL TRIAL: NCT05606367
Title: A Prospective, Randomized, Multicenter Clinical Trial of Non-slip Balloon Catheter in Patients With Coronary Artery Stenosis
Brief Title: Coronary Non-slip Balloon Catheter in Patients With Coronary Artery Stenosis(CREST)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAD-D-001
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Stenosis
Keywords: stenosis; coronary artery
MeSH Terms: conditions — Coronary Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-slip Balloon Catheter (Experimental): Subjects in experimental arm will be treated with the Non-slip Balloon Catheter manufactured by Shanghai Microport Rhythm Co. Ltd.
  Interventions: Device: Non-slip Balloon Catheter of Shanghai MicroPort Rhythm
- NSE Coronary Dilatation Catheter (Active Comparator): Subjects in control arm will be treated with Lacrosse® NSE manufactured by Goodman Medical Co. Ltd.
  Interventions: Device: NSE Coronary Dilatation Catheter

INTERVENTIONS:
Device: Non-slip Balloon Catheter of Shanghai MicroPort Rhythm — The principle of Non-slip Balloon Catheter in dilating stenotic lesions is mechanical extrusion of the vessel through the balloon, resulting in irregular rupture of atheromatous plaque and enlargement of the lumen.
  Arms: Non-slip Balloon Catheter
Device: NSE Coronary Dilatation Catheter — The Lacrosse® NSE is an angioplasty catheter with 3 longitudinal elements attached directly proximal and distal to the balloon that produces 3 endovascular surgical incisions during balloon dilation.
  Other Names: Lacrosse NSE
  Arms: NSE Coronary Dilatation Catheter

SUMMARY:
This is a prospective, multicenter, randomized controlled clinical investigation aiming to evaluate the safety and effectiveness of non-slip balloon catheter for the treatment of patients with coronary artery stenosis.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, randomized controlled clinical trial. 200 subjects are expected to be recruited in 7 research centers in China and randomly divided into two groups according to the ratio of test group: control group = 1:1. The primary endpoint is the acute lumen gain.

All subjects receive clinical follow-up during hospitalization and 30 days after surgery.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subjects aged≥18 years.
2. Subjects with silent myocardial ischemia, symptomatic angina pectoris, or old myocardial infarction.
3. Subjects who can undergo percutaneous coronary intervention (PCI).
4. Subjects who are able to understand the purpose of the trial, participate voluntarily and indicate by signing the informed consent form that they recognize the risks and benefits described in the informed consent document and are willing to undergo clinical follow-up.

Angiography Inclusion Criteria:

1. For subjects with single or double lesions, revascularization is required for up to two lesions; at most one non-target lesion can be treated in the same period, and the target lesion can be treated only after the treatment of non-target lesion meets the angiography success criteria and there is no complication. Target and non-target lesions must be located in different major epicardial vessels.
2. Target lesion meets criteria for revascularization:

   1. ≥ 70% and < 100% diameter stenosis; or
   2. ≥ 50% and < 70% diameter stenosis with clinical evidence of ischemia
3. Target lesion vessel diameter is between 2.0 mm and 4.0 mm (inclusive), target lesion length ≤ 30 mm.
4. Clinically judged to be the lesion that requires or is amenable to pretreatment with the study balloon catheter and that the study balloon catheter can pass after pre-dilatation.

General Exclusion Criteria:

1. Subjects who present with AMI recently (within 7 days).
2. Subjects who plan to undergo rotational atherectomy, laser coronary atherectomy, cutting balloon during target lesion pretreatment.
3. Subjects who are scheduled for PCI or CABG within 1 month of the index procedure.
4. Subjects with history of ischemic stroke or transient ischemic attack within 3 months.
5. Subjects with bleeding tendency, active gastrointestinal ulcer, history of cerebral hemorrhage or subarachnoid hemorrhage, contraindications to antiplatelet agents and anticoagulant therapy, and inability to receive antithrombotic therapy within 6 months.
6. Subjects who are scheduled for additional surgical procedures requiring discontinuation of aspirin, clopidogrel within 6 months of the baseline procedure.
7. Subjects with severe heart failure (NYHA III and above) or left ventricular ejection fraction(LVEF) < 35% (ultrasound or left ventriculography) and/or hemodynamic instability.
8. Subjects with unstable arrhythmias, such as high-risk premature ventricular contractions, ventricular tachycardia, high-grade atrioventricular block.
9. Subjects who are unable to receive antiplatelet therapy.
10. Subjects with hypersensitivity to aspirin, heparin, contrast agent, cobalt-based alloys (including metal elements such as cobalt, chromium, nickel, and tungsten), and polytetrafluoroethylene.
11. Subjects with renal insufficiency, serum creatinine greater than 177 μmol/L (2.0 mg/dl) or who are receiving hemodialysis.
12. Subjects who have been diagnosed with the terminal state of acute and chronic diseases such as advanced cancer and have a life expectancy of less than 1 year.
13. Subjects who have already received or are waiting for organ transplantation.
14. Subjects with blood routine test showed platelet count less than 50 × 10^9/L or more than 700 × 10^9/L, and/or hemoglobin less than 70 g/L.
15. Subjects who have participated in other clinical trials of drugs or medical devices before enrollment but have not been to the primary study endpoint until now.
16. Subjects who are judged by the investigator to be at high clinical risk for the use of the study device, unsuitable or non-compliant, and unable to complete the study as required.
17. Subjects who are pregnant or breastfeeding (women who may become pregnant must have a pregnancy test within 7 days prior to the baseline procedure).

Angiography Inclusion Criteria:

1. There are three severe lesions that needs revascularization.
2. Unprotected left main disease.
3. Target lesions meeting the following criteria:

   * Acute occlusion or thrombus;
   * Chronic total occlusion;
   * Bifurcation lesion;
   * Within 3 mm of the ostium of the left and right main coronary arteries (LAD/LCX/RCA);
   * CABG bridge stenosis;
   * Involved myocardial bridge;
   * Presence of dissection (Type C and above according to NHLBI classification);
   * Anatomy proximal to or within the target lesion that would preclude delivery of the study balloon catheter (e.g., severe tortuosity, etc.);
   * The study balloon catheter must pass previously implanted stent to reach target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Acute Lumen Gain | Baseline procedure
  Acute lumen gain is defined as the difference in the minimum lumen diameter of the target lesion before and after dilatation with the study balloon catheter (Microport or NSE Coronary Dilatation Catheter) as measured by QCA. (Acute lumen gain = minimum lumen diameter measured after dilatation with the study balloon catheter - minimum lumen diameter measured before dilatation with the study balloon catheter, AG=MLD post - MLD pre)

SECONDARY OUTCOMES:
Device success | Baseline procedure
  Device success is defined as successful delivery, inflation, deflation, and withdrawal of the study balloon catheter with < 50% diameter stenosis of the lesion after dilatation.
Lesion success | Baseline procedure
  Lesion success is defined as a target lesion with ≤ 30% residual stenosis and TIMI flow grade of 3 after treatment with any interventional method.
Procedural success | During hospitalization (up to 7 days after procedure)
  Procedure success is defined as having a target lesion with ≤ 30% diameter residual stenosis and TIMI flow grade of 3 after PCI procedure while the device was successful. There were no deaths, target vessel revascularization, or myocardial infarction during hospitalization (up to 7 days after baseline procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Bu, M.D., Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China